CLINICAL TRIAL: NCT01271777
Title: A Pilot Study to Evaluate the Efficacy of GFT505 (80mg) Orally Administered Once Daily for 8 Weeks on Insulin Sensitivity Using a Glucose Clamp Technique and Safety in Male Patients With Insulin Resistance and Abdominal Obesity. A Multicentre, Randomised, Single Blind, Placebo-Controlled, Cross Over Study.
Brief Title: Pilot Study With GFT505 (80mg) in Patients With Insulin Resistance and Abdominal Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GFT505-210-6; 2010-023219-32 (EudraCT Number)
Record Dates: First submitted 2011-01-04; First posted 2011-01-07 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Insulin Resistance; Abdominal Obesity
Keywords: Pre-diabetes; Clamp technique; PPARs; Insulin resistance
MeSH Terms: conditions — Insulin Resistance; Obesity, Abdominal; Glucose Intolerance | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GFT505 80mg (Experimental)
  Interventions: Drug: GFT505 80mg
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFT505 80mg — hard gelatin capsules dosed at 20mg, oral administration, 4 capsules per day before breakfast
  Arms: GFT505 80mg
Drug: Placebo — hard gelatin capsules, oral administration, 4 capsules per day before breakfast
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy on insulin sensitivity of GFT505 at 80mg/d in male patients with insulin resistance and abdominal obesity. Evaluation will be made using a glucose clamp technique.

DETAILED DESCRIPTION:
The study period per patient is 26 weeks: a selection period will precede a 8-week treatment period, a 6-week wash out period, a second 8-week treatment period in the second arm of treatment and a 2- week follow-up period.

Schedule:

* Selection visit prior to treatment period (D-14 and D-1)
* D0 : randomisation visit
* Period T1: first period of treatment with GFT505 80mg or placebo for 8 weeks (D1 to D56)
* Wash out period for 6 weeks (D57 to D98)
* Period T2: second period of treatment with GFT505 80mg or placebo for 8 weeks (D99 to D154)
* Follow up period for 2 weeks (D155 to D169)

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference ≥94cm.
* Body Mass Index ≤ 45kg/m2.
* Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) > 3.

Exclusion Criteria:

* Blood Pressure > 160 / 95 mmHg.
* Diabetes mellitus 1 or 2.
* Historical of bariatric surgery.
* Patient treated with a lipid-decreasing medication.
* A fasting plasma triglycerides concentration > 400mg/dL or a plasma Low Density Lipoprotein Cholesterol (LDL-c)concentration > 220mg/dL.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Glucose Infusion Rate (GIR) | 8 weeks
  To evaluate in each patient the differences in Glucose Infusion Rate (GIR) measured at the end of 8 weeks treatment periods with GFT505 (80 mg/day per os) or placebo according to a cross-over design.

SECONDARY OUTCOMES:
Differences in Hepatic Glucose Production (HGP) in each patient | 8 weeks
  To evaluate in each patient the differences in Hepatic Glucose Production (HGP) measured at the end of 8 weeks treatment periods with GFT505 (80 mg/day per os) or placebo according to a cross-over design.
Changes in GIR (Glucose Infusion Rate) | 8 weeks
  To compare the changes from baseline to endpoint in Glucose Infusion Rate (GIR). The baseline will be defined as the values of glucose clamp at V2. The same baseline will be used for the 2 periods. End-points will be defined as glucose clamp values at V4 for the first period and as glucose clamp values at V7 for the second period.
Changes in HGP (Hepatic Glucose Production) | 8 weeks
  To compare the changes from baseline to endpoint in Hepatic Glucose Production (HGP). The baseline will be defined as the values of glucose clamp at V2. The same baseline will be used for the 2 periods. End-points will be defined as glucose clamp values at V4 for the first period and as glucose clamp values at V7 for the second period.

CONTACTS AND LOCATIONS:
Overall Officials: Rémy Hanf, Development Director, Study Director — Genfit, France; Bertrand CARIOU, Pr., Study Chair — University Hospital of Nantes, France
Locations (2):
- France (2):
  - Site n°1, Nantes
  - Site n°2, Pierre-Bénite

REFERENCES:
- [Derived] Cariou B, Hanf R, Lambert-Porcheron S, Zair Y, Sauvinet V, Noel B, Flet L, Vidal H, Staels B, Laville M. Dual peroxisome proliferator-activated receptor alpha/delta agonist GFT505 improves hepatic and peripheral insulin sensitivity in abdominally obese subjects. Diabetes Care. 2013 Oct;36(10):2923-30. doi: 10.2337/dc12-2012. Epub 2013 May 28. PMID 23715754
- [Derived] Staels B, Rubenstrunk A, Noel B, Rigou G, Delataille P, Millatt LJ, Baron M, Lucas A, Tailleux A, Hum DW, Ratziu V, Cariou B, Hanf R. Hepatoprotective effects of the dual peroxisome proliferator-activated receptor alpha/delta agonist, GFT505, in rodent models of nonalcoholic fatty liver disease/nonalcoholic steatohepatitis. Hepatology. 2013 Dec;58(6):1941-52. doi: 10.1002/hep.26461. Epub 2013 Oct 29. PMID 23703580